CLINICAL TRIAL: NCT02220530
Title: Sedation Effect on the Global Quality Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hospital San Juan de Dios Tenerife (Other)
Responsible Party: Principal Investigator, Juan Salvador Baudet, Medical Doctor, Hospital San Juan de Dios Tenerife
Other Study IDs: HSJD-1
Record Dates: First submitted 2013-04-07; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Ambulatory Patients Referred for a First-time Colonoscopy
Keywords: Sedation.; Colonoscopy quality.; Scientific and technical quality.; Perceived quality (patient's satisfaction).; Safety
MeSH Terms: interventions — Conscious Sedation; Midazolam; Fentanyl

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sedation group: Colonoscopies performed with conscious sedation with iv midazolam and fentanyl
  Interventions: Drug: Conscious sedation with iv midazolam and fentanyl.
- Control group: Colonoscopies performed without sedation.

INTERVENTIONS:
Drug: Conscious sedation with iv midazolam and fentanyl. — Sedation group: Conscious sedation with iv midazolam and fentanyl dosed according to age, weight and baseline conditions of the patients.
  Other Names: Control group: Colonoscopies performed without sedation.
  Groups: Sedation group

SUMMARY:
This study aims to assess the impact of the use of sedation on the overall quality of the colonoscopy, therefore addressing each and every one of its dimensions, namely: scientific and technical quality, perceived quality and safety.

DETAILED DESCRIPTION:
In recent decades there has been a notable increase in the use of a range of gastrointestinal endoscopy procedures - colonoscopy particularly -, more so in recent years with the implementation of colorectal cancer screening programs.

Colonoscopy can cause discomfort and even pain. In order to reduce these effects and facilitate the procedure, patients are usually administered iv sedation.

Numerous studies have assessed the impact of sedation on patient discomfort and anxiety, on the undesirable effects of the colonoscopy, and even on certain aspects relating to its scientific and technical quality. There have not, however, been any studies evaluating the effects of sedation on the overall quality of the procedure.

The overall quality of every medical act can be defined according to four dimensions: accessibility, or how easily the patient can obtain the assistance required without physical or bureaucratic barriers; scientific and technical quality, or the provision of the best possible assistance with the most up-to-date knowledge and technical resources; perceived quality, or the patient's degree of satisfaction with the care provided; and safety, or the absence of undesirable side effects. Doctors have typically assessed the quality of a procedure based on its scientific and technical quality and its safety. The investigators have strived to conduct good, complication-free techniques based on cutting-edge scientific knowledge, but have often overlooked the other dimensions.

This study aims to assess the impact of the use of sedation on the overall quality of the colonoscopy, therefore addressing each and every one of its dimensions, namely: scientific and technical quality, perceived quality and safety. Since sedation during the procedure has no impact on accessibility, the study will not assess this dimension.

Subjects and Methods:

Prospective case-control study. The study will include consecutive ambulatory patients referred to our Endoscopy Unit for a first-time colonoscopy. Patients will be excluded when they have had previous colonoscopies, have an anesthetic risk above ASA III (American Society of Anesthesia classifications) allergy to the drugs used or if they are undergoing antiplatelet or anticoagulant therapy contraindicated for the procedure, pregnant woman and patients unable to understand the questionnaires.

Prior to inclusion demographic data, clinical background and indication for the colonoscopy will be collected on each patient.

Thereafter patients will be randomly assigned to colonoscopy without sedation or with conscious sedation with iv midazolam and fentanyl dosed according to age, weight and baseline conditions.

The procedures will be conducted by four endoscopists with ample experience in endoscopy and sedation (over 7000 colonoscopies each).

1. Data collected during the endoscopy will include:

   1. The degree of cleanliness of the colon according to the Boston scale; defined as the adequate preparation of at least 2 points in each region of the colon);
   2. Whether or not colonoscopy is completed up to the cecum;
   3. Time needed for insertion up to the cecum and for withdrawal;
   4. The complications that might arise during the procedure and recovery period (early complications). To this end, patients' oxygen saturation and heart rate will be continuously monitored from the beginning of the procedure until their discharged and their blood pressure will be taken every 5 minutes. Non-sedated patients will be discharged from the Unit immediately after the procedure, and sedated patients when they reach a score of 9 or 10 on the Aldrete scale.
   5. Adenomas resected, based on pathology reports. All of the biopsies will be examined by a pathologist specialized in gastrointestinal pathology.
2. Thirty days after the Endoscopy, patients will be interviewed by telephone by staff with no involvement in the study (call center) and asked to respond to two questionnaires.

   1. The ASGE (American Society of Gastrointestinal Endoscopy) endoscopy satisfaction survey (GHAA 9-me), previously translated into Spanish and validated by our team.
   2. A survey on complications suffered in the 30 days following the procedure (late complications), previously used in earlier studies.
3. Assessment of quality criteria:

   1. Six indicators will be used to assess the scientific and technical quality of each procedure. The first three will assess their technical aspects: percentage of colonoscopies completed up to the cecum; time required to reach the cecum; and withdrawal time. The remaining three are results indicators: percentage of patients with adenomas; total number of adenomas per patient; and total number of advanced adenomas. These indicators were previously validated in our setting.

      Since the use or not of sedation during the procedure does not affect the cleanliness of the colon, this indicator will be used as a control variable.
   2. Perceived quality will be assessed using the ASGE (American Society of Gastrointestinal Endoscopy) satisfaction survey, previously translated into Spanish and adapted and validated. Total scores, scores for the procedure (item 7 on the survey) and the number of patients rating the procedure "excellent" will be analyzed.
   3. Safety will be assessed following the same method used in previous research, analyzing early complications (those occurring during the procedure and recovery phase) and late complications (those occurring in the 30 days after the procedure).

Statistical Analyses:

Results will be expressed as mean ± standard deviation. Comparisons between groups will be performed using the Chi-squared test for ordinal variables and Student's t-test for quantitative variables. Results with a p value <0.05 will be considered statistically significant. Logistic regression will be used to determine the impact of sedation on the quality indicators studied.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive ambulatory patients referred to our Endoscopy Unit for a first-time colonoscopy.

Exclusion Criteria:

* Patients with previous colonoscopies.
* Patients with anesthetic risk above ASA III,
* Patients with allergy to the drugs used.
* Patients undergoing antiplatelet or anticoagulant therapy.
* Pregnant woman.
* Patients unable to understand the questionnaires.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective case-control study. The study will include . Patients will be excluded when they have had previous colonoscopies, have an anesthetic risk above ASA III, allergy to the drugs used or if they are undergoing antiplatelet or anticoagulant therapy contraindicated for the procedure
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of colonoscopies completed up to the cecum. | During colonoscopy
  Colonoscopy in which the cecum is reached per hundred colonoscopy performed
Time required to reach the cecum | During colonoscopy
  Time used to complete colonoscopy (in minutes)
Endoscopic withdrawal time | During colonoscopy
  Time used (in minutes) to endoscopic withdrawal.
Adenomas resected | During colonoscopy
  Number of adenomas resected
Perceived quality (patients satisfaction). | Thirty days after colonoscopy
  ASGE (American Society of Gastrointestinal Endoscopy) endoscopy satisfaction survery score (GHAA 9-me).
Early complications. | During colonoscopy.
  Complications occurring during the procedure and recovery phase.
Late complications. | Thirty days after colonoscopy
  Complications occurring in the 30 days after the procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Salvador Baudet, M. D., Principal Investigator — Hospital San Juan de Dios Tenerife
Locations (1):
- Htal. Universitario Ntra. Sra. de Candelaria, Santa Cruz de Tenerife, Santa Cruz de Tenerife, Spain

REFERENCES:
- [Background] Gellad ZF, Weiss DG, Ahnen DJ, Lieberman DA, Jackson GL, Provenzale D. Colonoscopy withdrawal time and risk of neoplasia at 5 years: results from VA Cooperative Studies Program 380. Am J Gastroenterol. 2010 Aug;105(8):1746-52. doi: 10.1038/ajg.2010.107. Epub 2010 Mar 16. PMID 20234348
- [Background] Bannert C, Reinhart K, Dunkler D, Trauner M, Renner F, Knoflach P, Ferlitsch A, Weiss W, Ferlitsch M. Sedation in screening colonoscopy: impact on quality indicators and complications. Am J Gastroenterol. 2012 Dec;107(12):1837-48. doi: 10.1038/ajg.2012.347. Epub 2012 Nov 13. PMID 23147522
- [Background] Rex DK, Petrini JL, Baron TH, Chak A, Cohen J, Deal SE, Hoffman B, Jacobson BC, Mergener K, Petersen BT, Safdi MA, Faigel DO, Pike IM; ASGE/ACG Taskforce on Quality in Endoscopy. Quality indicators for colonoscopy. Am J Gastroenterol. 2006 Apr;101(4):873-85. doi: 10.1111/j.1572-0241.2006.00673.x. No abstract available. PMID 16635231
- [Background] Rex DK. Quality in colonoscopy: cecal intubation first, then what? Am J Gastroenterol. 2006 Apr;101(4):732-4. doi: 10.1111/j.1572-0241.2006.00483.x. PMID 16635220
- [Background] Baudet JS, Aguirre-Jaime A. The sedation increases the acceptance of repeat colonoscopies. Eur J Gastroenterol Hepatol. 2012 Jul;24(7):775-80. doi: 10.1097/MEG.0b013e32835376a2. PMID 22522140
- [Background] Sanchez Del Rio A, Baudet JS, Naranjo Rodriguez A, Campo Fernandez de Los Rios R, Salces Franco I, Aparicio Tormo JR, Sanchez Munoz D, Llach J, Hervas Molina A, Parra-Blanco A, Diaz Acosta JA; los miembros del Grupo de Calidad en Endoscopia de la Asociacion Espanola de Gastroenterologia. [Development and validation of quality standards for colonoscopy]. Med Clin (Barc). 2010 Jan 30;134(2):49-56. doi: 10.1016/j.medcli.2009.07.047. Epub 2009 Nov 14. Spanish. PMID 19913837
- [Background] Baudet JS, Borque P, Borja E, Alarcon-Fernandez O, Sanchez-del-Rio A, Campo R, Aviles J. Use of sedation in gastrointestinal endoscopy: a nationwide survey in Spain. Eur J Gastroenterol Hepatol. 2009 Aug;21(8):882-8. doi: 10.1097/MEG.0b013e328314b7ca. PMID 19352194
- [Background] Baudet JS, Diaz-Bethencourt D, Aviles J, Aguirre-Jaime A. Minor adverse events of colonoscopy on ambulatory patients: the impact of moderate sedation. Eur J Gastroenterol Hepatol. 2009 Jun;21(6):656-61. doi: 10.1097/MEG.0b013e328314b7e3. PMID 19300274
- [Background] Del Rio AS, Baudet JS, Fernandez OA, Morales I, Socas Mdel R. Evaluation of patient satisfaction in gastrointestinal endoscopy. Eur J Gastroenterol Hepatol. 2007 Oct;19(10):896-900. doi: 10.1097/MEG.0b013e3281532bae. PMID 17873615
- [Background] Sanchez del Rio A, Alarcon Fernandez O, Baudet JS, Sainz Menendez Z, Socas Mendez M. Reliability of the Spanish version of a brief questionnaire on patient satisfaction with gastrointestinal endoscopy. Rev Esp Enferm Dig. 2005 Aug;97(8):554-61. doi: 10.4321/s1130-01082005000800003. English, Spanish. PMID 16266222
- [Background] Kahi CJ, Ballard D, Shah AS, Mears R, Johnson CS. Impact of a quarterly report card on colonoscopy quality measures. Gastrointest Endosc. 2013 Jun;77(6):925-31. doi: 10.1016/j.gie.2013.01.012. Epub 2013 Mar 6. PMID 23472996
- [Background] Valori R, Rey JF, Atkin WS, Bretthauer M, Senore C, Hoff G, Kuipers EJ, Altenhofen L, Lambert R, Minoli G; International Agency for Research on Cancer. European guidelines for quality assurance in colorectal cancer screening and diagnosis. First Edition--Quality assurance in endoscopy in colorectal cancer screening and diagnosis. Endoscopy. 2012 Sep;44 Suppl 3:SE88-105. doi: 10.1055/s-0032-1309795. Epub 2012 Sep 25. PMID 23012124
- [Background] Williams JE, Holub JL, Faigel DO. Polypectomy rate is a valid quality measure for colonoscopy: results from a national endoscopy database. Gastrointest Endosc. 2012 Mar;75(3):576-82. doi: 10.1016/j.gie.2011.12.012. PMID 22341104
- [Background] Lee TJ, Rutter MD, Blanks RG, Moss SM, Goddard AF, Chilton A, Nickerson C, McNally RJ, Patnick J, Rees CJ. Colonoscopy quality measures: experience from the NHS Bowel Cancer Screening Programme. Gut. 2012 Jul;61(7):1050-7. doi: 10.1136/gutjnl-2011-300651. Epub 2011 Sep 22. PMID 21940723
- [Background] Imperiali G, Minoli G, Meucci GM, Spinzi G, Strocchi E, Terruzzi V, Radaelli F. Effectiveness of a continuous quality improvement program on colonoscopy practice. Endoscopy. 2007 Apr;39(4):314-8. doi: 10.1055/s-2006-945196. Epub 2007 Feb 1. PMID 17273959